CLINICAL TRIAL: NCT06649565
Title: Prospective Validation and Application of an Artificial Intelligence-based Model for Evaluating the Efficacy of Breast Cancer Patients After Neoadjuvant Therapy
Status: Recruiting | Type: Observational
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, PENG YUAN, Chief Physician, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Other Study IDs: 2024-1- 4021
Record Dates: First submitted 2024-06-24; First posted 2024-10-18 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-08

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Breast cancer patients who achieved pathological complete response after neoadjuvant therapy: All enrolled breast cancer patients received normal neoadjuvant therapy and subsequent surgery without intervention in the diagnosis and treatment process. They were judged to have achieved pathological complete respone based on surgical pathology.
  Interventions: Other: no intervention
- Breast cancer patients who did not achieve pathological complete response after neoadjuvant therapy: All enrolled breast cancer patients received normal neoadjuvant therapy and subsequent surgery without intervention in the diagnosis and treatment process. They were judged as not achieving pathological complete respone based on surgical pathology.
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
Breast cancer has become the world's number one cancer. While its therapeutic efficacy is increasing, how to achieve non-invasive evaluation of the efficacy of neoadjuvant therapy (NAT) for breast cancer patients and thus avoid surgery has become a bottleneck problem that needs to be broken through in clinical diagnosis and treatment. Existing non-invasive evaluation strategies are limited to single-center, single-modality modeling, and have problems such as low performance and poor versatility. Therefore, in the early stage of this study, multi-modality breast cancer patient data from multiple centers across the country were collected and the establishment of an artificial intelligence (AI) efficacy prediction model was preliminarily completed. On this basis, this project intends to further improve the multi-center prospective validation study of the prediction model. The research results will help solve the scientific problem of non-invasive judgment of NAT efficacy in breast cancer patients and provide a new paradigm for the research of high-performance AI diagnosis and treatment auxiliary systems applicable to multiple centers.

DETAILED DESCRIPTION:
(1) Prospectively collect breast MRI original images (DCE and ADC sequences) and corresponding clinical and surgical pathological data of multi-center breast cancer patients before and after neoadjuvant treatment, store and transport them via mobile hard disks, and input the processed data into the established efficacy determination model stored in a dedicated cloud server; (2) Use artificial intelligence to automatically delineate the ROI area and extract the imaging genomics and deep learning features therein, and combine the clinical pathological characteristics of the patients to further prospectively verify the effectiveness of the established pCR efficacy determination model.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were treated in the above research centers between January 1, 2024 and October 31, 2025;
* ≥18 years old, female, ECOG score ≤2;
* Pathological biopsy confirmed invasive breast cancer;
* AJCC (8th edition) stage I-III;
* MRI imaging data before and after neoadjuvant therapy;
* Planned mastectomy or breast-conserving surgery after neoadjuvant therapy, and postoperative pathological information obtained.

Exclusion Criteria:

* Bilateral breast cancer, multiple lesions, or occult breast cancer;
* Poor MRI data quality;
* Patients who had received other anti-tumor treatments before enrollment;
* Patients with other malignant tumors

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study adopts sequential enrollment (continuously recruiting patients until the sample size requirement is met). The subjects are patients with neoadjuvant treatment for breast cancer who were treated in Beijing Second Hospital, Beijing Luhe Hospital Affiliated to Capital Medical University, and Beijing Sanhuan Cancer Hospital from January 2024 to December 2026. Each independent medical center will include 100 patients, for a total of 300 patients.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Breast MRI radiomics characteristics of breast cancer patients during neoadjuvant therapy | Breast cancer MRI images before neoadjuvant therapy and immediately after completing neoadjuvant therapy

CONTACTS AND LOCATIONS:
Overall Officials: peng yuan, doctor, Study Director — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (2):
- China (2):
  - Sanhuan Cancer Hospital, Chaoyang District, Beijing(Cancer Hospital, Chinese Academy of Medical Sciences, close medical alliance), Beijing, Beijing Municipality
  - Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: No